CLINICAL TRIAL: NCT00469092
Title: A Multi-national, Open-labelled, Randomised, Parallel Group, 4 Week run-in and 26 Weeks Treat-to-target Comparison of Biphasic Insulin Aspart 30 Once Daily Versus Insulin Glargine Once Daily Both in Combination With Metformin and Glimepiride in Insulin naïve Subjects With Type 2 Diabetes
Brief Title: Comparison of Biphasic Insulin Aspart 30 Versus Insulin Glargine Both in Combination With Metformin and Glimepiride in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1731; 2006-003288-29 (EudraCT Number)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Glargine; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart; Drug: metformin; Drug: glimepiride
- Glargine (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: metformin; Drug: glimepiride

INTERVENTIONS:
Drug: biphasic insulin aspart — Treat-to-target dose titration scheme. The titration scheme is based on the previous 3 days fasting plasma glucose (FPG) measurements.
  Arms: BIAsp 30
Drug: insulin glargine — Treat-to-target dose titration scheme. The titration scheme is based on the previous 3 days fasting plasma glucose (FPG) measurements.
  Arms: Glargine
Drug: metformin — Tablets, 2550 mcg. Administered once daily.
Drug: glimepiride — Tablets 2 mg. 4, 6 or 8 mg administered once daily.

SUMMARY:
This trial is conducted in Africa, Asia, Europe, Oceania and South America.

This trial aims for a comparison of biphasic insulin aspart 30 once daily versus insulin glargine once daily all in combination with metformin and glimepiride in insulin naive subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treatment with OADs (Oral Anti-Diabetic Drugs) for more than 6 months
* Ongoing stable treatment with metformin for at least 2 months
* Ongoing stable treatment with minimum half maximal dose of any insulin secretagogue for at least 2 months
* Insulin naive
* HbA1c (glycosylated haemoglobin A1c) between 7.0% and 11.0% (inclusive of both values)

Exclusion Criteria:

* Metformin contraindication according to local practice
* TZD (thiazolidinedione) treatment for the last 5 months before trial start
* Systemic treatment with any corticosteroid 3 months before trial start
* Any disease or condition which according to the Investigator would interfere with the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (65):
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad Autonoma de Bs As
  - Novo Nordisk Investigational Site, Ciudad Autónoma de BsAs
  - Novo Nordisk Investigational Site, Mar del Plata
- Austria (5):
  - Novo Nordisk Investigational Site, Bregenz
  - Novo Nordisk Investigational Site, Feldkirch
  - Novo Nordisk Investigational Site, Traisen
  - Novo Nordisk Investigational Site, Vienna
  - Novo Nordisk Investigational Site, Wels
- Czechia (2):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Hradec Králové
- France (6):
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Limoges
  - Novo Nordisk Investigational Site, Mougins
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Pointe à Pitre
- India (4):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Karnāl, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Visakhapatnam
- Malaysia (3):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Pulau Pinang
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Pachuca
- Netherlands (5):
  - Novo Nordisk Investigational Site, Almere Stad
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Leiderdorp
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Zoetermeer
- Philippines (2):
  - Novo Nordisk Investigational Site, Manila
  - Novo Nordisk Investigational Site, Quezon City
- Poland (14):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Gdynia
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lubin
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Olsztyn
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Rzeszów
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Romania (5):
  - Novo Nordisk Investigational Site, Satu Mare, Satu Mare County
  - Novo Nordisk Investigational Site, Botoșani
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Galati
  - Novo Nordisk Investigational Site, Târgovişte
- Serbia and Montenegro (3):
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Nis
  - Novo Nordisk Investigational Site, Novi Sad
- South Africa (3):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
- Spain (3):
  - Novo Nordisk Investigational Site, Alzira
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
- Sweden (4):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm

REFERENCES:
- [Result] Strojek K, Bebakar WM, Khutsoane DT, Pesic M, Smahelova A, Thomsen HF, Kalra S. Once-daily initiation with biphasic insulin aspart 30 versus insulin glargine in patients with type 2 diabetes inadequately controlled with oral drugs: an open-label, multinational RCT. Curr Med Res Opin. 2009 Dec;25(12):2887-94. doi: 10.1185/03007990903354674. PMID 19821654
- [Result] Kalra S, Plata-Que T, Kumar D, Mumtaz M, Sondergaard F, Kozlovski P, Bebakar WM. Initiation with once-daily BIAsp 30 results in superior outcome compared to insulin glargine in Asians with type 2 diabetes inadequately controlled by oral anti-diabetic drugs. Diabetes Res Clin Pract. 2010 Jun;88(3):282-8. doi: 10.1016/j.diabres.2010.03.004. Epub 2010 Apr 2. PMID 20363044
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled 64 sites in 15 countries in Africa, Europe, Asia, North America and South America.
Pre-assignment Details: A screening period of 1-2 weeks was followed by a run-in period of 4 weeks during which metformin was titrated to maximum 2550 mg and glimepiride to 4 mg, at the discretion of the investigator. Subjects who were already taking 4, 6 or 8 mg glimepiride continued on this dose. Doses were kept constant during the last week prior to randomisation.
Groups:
- BIAsp 30: Biphasic insulin aspart 30 + metformin + glimepiride
- Glargine: Insulin glargine + metformin + glimepiride
Period: Overall Study
Arm/Group | BIAsp 30 | Glargine
Started | 239 | 241
Exposed to Study Drug | 231 | 238
Completed | 213 | 220
Not Completed | 26 | 21
Not completed — Adverse Event | 5 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Withdrawal Criteria | 3 | 4
Not completed — Incorrectly Randomised | 4 | 3
Not completed — Contraindication metformin/glimepiride | 1 | 0
Not completed — Use of lipid lowering drug | 1 | 0
Not completed — Hypoglycaemic Episodes | 1 | 1
Not completed — Abnormal lab value | 1 | 0
Not completed — Use of Corticosteroid | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIAsp 30 | Glargine | Total
Number analyzed (Participants) | 231 | 238 | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (9.7) | 56.1 (10.0) | 56.0 (9.9)
Gender [Count of Participants; unit: Participants]
  Female | 123 | 140 | 263
  Male | 108 | 98 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 40 | 75
  Not Hispanic or Latino | 192 | 196 | 388
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 11 | 24
  Asian | 76 | 79 | 155
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 7 | 17
  White | 125 | 133 | 258
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 4 | 2 | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 29.0 (4.6) | 29.1 (4.6) | 29.1 (4.6)
Diabetes duration [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of diabetes
  years | 9.1 (5.8) | 9.5 (6.1) | 9.3 (6.0)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated Haemoglobin
  percentage of total haemoglobin | 8.9 (1.0) | 9.0 (1.1) | 9.0 (1.1)
Weight [Mean (Standard Deviation); unit: kg] | 77.5 (14.6) | 77.3 (15.4) | 77.4 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Glycosylated Haemoglobin A1c measured in blood samples after 26 weeks of treatment.
Time Frame: After 26 weeks of treatment
Population: Intention to Treat (Last Observation Carried Forward) population. All randomised subjects exposed to trial drug, and who had at least a baseline HbA1c measurement and at least one post randomisation HbA1c measurement.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of total haemoglobin
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 225 | 232
percentage of total haemoglobin | 7.08 (0.07) | 7.23 (0.07)
Statistical Analysis 1: Comparison: BIAsp 30 vs Glargine; HbA1c was compared between the treatment groups by fitting a linear regression model (ANCOVA) with treatment and country as factors and the baseline values as a continuous covariate. Mean and SE are estimated from the model; Test type: Non-Inferiority or Equivalence — Non-inferiority is shown if the upper limit of the 95% CI is less than 0.4%. Furthermore, superiority of BIAsp 30 OD over insulin glargine OD was shown if the upper limit of the 95% CI for the difference is lower than 0%. Equivalence is shown if the upper limit of the 95% CI for the difference is lower than 0.4% and the lower limit of the 95% CI is greater than -0.4%; p = 0.029, Regression, Linear — P-value is for the test for difference in means equals 0 against the alternative that the difference is different from 0; Mean Difference (Net) = -0.16, 95% CI [-0.30 to -0.02]

2. Secondary Outcome: 9-point Self-measured Plasma Glucose Profiles
Description: Glycaemic control measured by 9-point self-measured plasma glucose (SMPG) profiles. The 9 time points for self-measurement during the day were: Before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, before bedtime, at 2-4 AM, and before breakfast the following day. Hypoglycaemia episodes were defined as major or minor. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L or 56 mg/dL.
Time Frame: After 26 weeks of treatment
Population: Intention to Treat, Last Observation Carried Forward population. All randomised subjects exposed to trial drug, and who had at least a baseline HbA1c measurement and at least one post randomisation HbA1c measurement.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 225 | 232
mmol/L
  Before breakfast | 6.73 (0.12) | 6.56 (0.12)
  2 hours after breakfast | 9.40 (0.20) | 9.07 (0.20)
  Before lunch | 7.24 (0.18) | 7.28 (0.18)
  2 hours after lunch | 8.90 (0.20) | 8.98 (0.20)
  Before dinner | 7.90 (0.18) | 7.80 (0.18)
  2 hours after dinner | 8.66 (0.19) | 9.18 (0.19)
  Before bedtime | 7.77 (0.18) | 8.54 (0.18)
  02:00-04:00 AM | 6.56 (0.14) | 6.69 (0.14)
  Before breakfast following day | 6.65 (0.12) | 6.40 (0.12)
Statistical Analysis 1: Comparison: BIAsp 30 vs Glargine; The profiles were compared between the treatment groups by fitting a repeated measures mixed model including treatment, time, the treatment-by-time interaction and country as fixed effects, and subject as random effect; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis — P-value for parallelism is overall test for parallel time profiles between treatment groups i.e. time by treatment group interaction effect

3. Secondary Outcome: Number of Subjects Achieving the Treatment Target for Glycosylated Haemoglobin A1c (HbA1c)
Description: The number of subjects achieving the treatment target for glycosylated haemoglobin A1c after 26 weeks treatment. The treatment targets were: HbA1c <= 6.5% of haemoglobin and HbA1c < 7% of haemoglobin.
Time Frame: After 26 weeks of treatment
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 225 | 232
participants
  HbA1c <= 6.5% of haemoglobin | 54 | 60
  HbA1c < 7.0% of haemoglobin | 101 | 106
  Reduction > 1% point from baseline | 134 | 132
  HbA1c < 7% no nocturnal hypoglycemia | 82 | 92
  HbA1c < 7%, no daytime hypoglycemia | 52 | 50
  HbA1c < 7%, no hypoglycemia | 45 | 45
Statistical Analysis 1: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 0.914, 95% CI [0.57 to 1.47] — The OR and 95% CI is for the HbA1c <= 6.5% treatment target
Statistical Analysis 2: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 1.014, 95% CI [0.67 to 1.54] — The OR and 95% CI is for the HbA1c < 7.0% treatment target
Statistical Analysis 3: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 1.131, 95% CI [0.72 to 1.77] — The OR and 95% CI is for the reduction more than 1.0% from baseline treatment target
Statistical Analysis 4: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 0.905, 95% CI [0.59 to 1.38] — The OR and 95% CI is for the HbA1c < 7% no nocturnal (00:00-06:00) hypoglycemia treatment target
Statistical Analysis 5: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 1.181, 95% CI [0.74 to 1.87] — The OR and 95% CI is for the HbA1c < 7%, no daytime (06:01-23:59) hypoglycemia treatment target
Statistical Analysis 6: Comparison: BIAsp 30 vs Glargine; Test type: Superiority or Other; Odds Ratio (OR) = 1.122, 95% CI [0.69 to 1.82] — The OR and 95% CI is for the HbA1c < 7%, no hypoglycemia treatment target

4. Secondary Outcome: Treatment Satisfaction as Measured by the Diabetes Medication Satisfaction Questionnaire (Diab MedSat)
Description: Subjects assessed the burden, efficacy, symptoms and overall score in the treatment satisfaction questionnaire, Diab MedSat (Diabetes Medication Satisfaction questionnaire). The scores were transformed to a 0-100 scale with higher scores indicating greater satisfaction. The score of the subscales was computed as the mean of the items in each subscale.
Time Frame: After 26 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 225 | 232
scores on a scale
  Burden Score | 83.10 (1.13) | 83.06 (1.16)
  Efficacy Score | 73.25 (1.57) | 73.47 (1.57)
  Symptoms Score | 72.42 (1.29) | 72.81 (1.29)
  Overall Score | 76.53 (1.04) | 76.64 (1.05)
Statistical Analysis 1: Comparison: BIAsp 30 vs Glargine; The Diab MedSat measure was scored as an overall score as well as three subscale scores. The scores were transformed to a 0-100 scale with higher scores indicating greater satisfaction. The score of the subscales was computed as the mean of the items in each subscale. The overall score is the mean of all three subscales; Test type: Superiority or Other; Mean Difference (Net) = 0.04, 95% CI [-2.40 to 2.48] — The mean difference and 95% CI is for the burden score. The scores were compared between the treatment groups by fitting a linear regression model with treatment and country as factors and the baseline values as a continuous covariate
Statistical Analysis 2: Comparison: BIAsp 30 vs Glargine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -0.22, 95% CI [-3.56 to 3.11] — The mean difference and 95% CI is for the efficacy score. The scores were compared between the treatment groups by fitting a linear regression model with treatment and country as factors and the baseline values as a continuous covariate
Statistical Analysis 3: Comparison: BIAsp 30 vs Glargine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Net) = -0.39, 95% CI [-3.14 to 2.35] — The mean difference and 95% CI is for the symptoms score. The scores were compared between the treatment groups by fitting a linear regression model with treatment and country as factors and the baseline values as a continuous covariate
Statistical Analysis 4: Comparison: BIAsp 30 vs Glargine; Diab MedSat measure was scored as an overall score as well as three subscale scores, and transformed to a 0-100 scale with higher scores indicating greater satisfaction. The score of the subscales was computed as the mean of the items in each subscale. The overall score is the mean of all three subscales; Test type: Superiority or Other; Regression, Linear; Mean Difference (Net) = -0.11, 95% CI [-2.36 to 2.14] — The mean difference and 95% CI is for the overall score. The scores were compared between the treatment groups by fitting a linear regression model with treatment and country as factors and the baseline values as a continuous covariate

5. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes experienced in each treatment arm. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L or 56 mg/dL. Symptoms only if subject was able to treat her/himself and with either no plasma glucose or blood glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L or 56 mg/dL.
Time Frame: Weeks 0-26
Measure: Number; unit: events
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 231 | 238
events
  Minor | 443 | 318
  Symptom only | 265 | 224
  Major | 3 | 3
  Unclassified | 1 | 0

6. Secondary Outcome: Number of Subjects Reporting Treatment Emergent Adverse Events
Description: Number of subjects reporting treatment emergent adverse events during the trial (from week 0 to week 26). Adverse events were reported as treatment emergent if they occurred from the date of first insulin trial product administration up to and including the date of last insulin trial product administration.
Time Frame: Weeks 0-26
Population: The safety analysis population consists of all subjects exposed to trial products.
Measure: Number; unit: participants
Arm/Group | BIAsp 30 | Glargine
Number analyzed (Participants) | 231 | 238
participants | 117 | 115

ADVERSE EVENTS:
Time Frame: The adverse event were collected in a time span of 26 weeks.
Description: The safety analysis population consists of all subjects exposed to trial products.
Arm/Group | BIAsp 30 | Glargine
Serious Adverse Events (participants affected / at risk) | 13/231 | 10/238
Other Adverse Events (participants affected / at risk) | 56/231 | 63/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=231) | Glargine (N=238)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 (1) | 0 (0)
Otitis Media Chronic (Infections and infestations) | 1 (1) | 0 (0)
Perianal Abscess (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Primary Atypical (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic Foot (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemic Unconsciousness (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 2 (2)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic Coma (Nervous system disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wart Excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Arterial Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (2)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=231) | Glargine (N=238)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 13 (14)
Nasopharyngitis (Infections and infestations) | 20 (22) | 20 (23)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (12) | 14 (20)
Headache (Nervous system disorders) | 18 (29) | 16 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any plans for publications and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.